CLINICAL TRIAL: NCT01324102
Title: Yoga Cancer Rehabilitation Study
Brief Title: Yoga Cancer Rehabilitation Study: A Randomized Trial of Adaptive Yoga for Older Cancer Survivors
Acronym: YogaCares
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7629-P
Record Dates: First submitted 2011-03-04; First posted 2011-03-28 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Neoplasms
Keywords: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Yoga therapy (Active Comparator): The intervention is an 8 week Yoga therapy class adapted to the specific needs of the veteran. The class meets two times per weeks for 90 minutes. A series of poses are instructed, with adaptations used as provided by a physical therapist.
  Interventions: Behavioral: Yoga therapy
- 2. Wait list (No Intervention): The comparative intervention is an 8 week wait list control group for which there is no intervention provided within the study protocol.

INTERVENTIONS:
Behavioral: Yoga therapy — For the second aim of the study, individuals will complete an 8 week yoga intervention in a non-randomized trial to establish safe procedures for yoga for an older post colorectal cancer veteran population.
  Arms: 1. Yoga therapy

SUMMARY:
With advances in the detection and treatment of cancer, there are now 14 million cancer survivors in the U.S., 500,000 of whom are treated in the Veterans Health Administration. The mental and physical health consequences of cancer and its treatment may affect a Veteran's functioning and re-integration back into family, work, and daily life. Recent studies suggest that yoga may be an effective intervention for improving both the physical and mental health of individuals after cancer, although this has not been studied in Veterans. This study has three components: (1) Determine factors that increase participation in Yoga by Veterans using individual interviews and focus group; (2) Create a Yoga protocol for Veterans adapted from an existing empirically supported treatment, akin to a phase 1 clinical trial for safety and tolerability; (3) Evaluate the efficacy of Yoga for improving fatigue, insomnia, anxiety, and depression after treatment for colorectal cancer, akin to a phase 2 trial with randomization.

DETAILED DESCRIPTION:
With a 1 and 2 lifetime risk of diagnosis, cancer is a highly prevalent disease. Cancer and its treatment are associated with long term mental and physical side effects that impair physical, vocational, and social role functioning. In order to provide excellent care for Veterans, rehabilitative strategies to improve mental and physical health after cancer treatment need empirical study. The objective of the proposed pilot project is to create a Veterans' Yoga Rehabilitation Program for cancer survivors who receive care in the Veterans Health Administration, that is based on an existing evidence based protocol which is systemically adapted, marketed, and tested in a Veteran population, with 3 aims:

Aim 1: Enhancing Acceptability To determine factors that will increase participation in Yoga in Veterans after treatment for cancer, who are primarily male and older than age 60.

Aim 2: Adapting to Veterans To create a Yoga protocol by adapting an empirically supported Yoga protocol to the needs of Veterans.

Aim 3: Evaluating Efficacy To evaluate the efficacy of the Yoga protocol for improving health related quality of life in four domains, and, to determine if efficacy varies as a function of patient age or pre-existing Post Traumatic Stress Disorder. The long term goal is to develop an evidence based mind-body Yoga intervention to support healing and restore function in Veterans Health Administration patients for use after treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Cancer treated in the past 3 years

Exclusion Criteria:

* Dementia
* Psychotic Disorder
* In hospice care

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ann Moye, PhD, Principal Investigator — VA Boston Healthcare System Brockton Campus, Brockton, MA
Locations (1):
- VA Boston Healthcare System Brockton Campus, Brockton, MA, Brockton, Massachusetts, United States

REFERENCES:
- [Background] Culos-Reed SN, Carlson LE, Daroux LM, Hately-Aldous S. A pilot study of yoga for breast cancer survivors: physical and psychological benefits. Psychooncology. 2006 Oct;15(10):891-7. doi: 10.1002/pon.1021. PMID 16374892
- [Background] Danhauer SC, Tooze JA, Farmer DF, Campbell CR, McQuellon RP, Barrett R, Miller BE. Restorative yoga for women with ovarian or breast cancer: findings from a pilot study. J Soc Integr Oncol. 2008 Spring;6(2):47-58. PMID 18544284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants identified through cancer registry who were: diagnosed with cancer (any type) Stage 1-4 within the past three years; received surgery, chemotherapy, or radiation treatment; no psychotic or dementing disorders; and not currently in hospice care.
Pre-assignment Details: No participants were excluded prior to assignment.
Groups:
- Yoga Therapy Intervention: Intervention
  Yoga therapy received an 8 week 2x weekly Yoga therapy class.
- Wait List Control: Wait List control received no intervention for 8 weeks, then joined the yoga group
Period: Overall Study
Arm/Group | Yoga Therapy Intervention | Wait List Control
Started | 11 (Yoga groups 3 and 5 (not including pre-randomization group)) | 12 (Yoga group 4 and 6)
Completed | 10 | 6
Not Completed | 1 | 6
Not completed — illness | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Yoga Therapy Intervention: Intervention: Yoga therapy was 8 week class for two times per week
- Wait List Control: Wait List control: The wait list control did not receive an intervention.
- Total: Total of all reporting groups
Arm/Group | Yoga Therapy Intervention | Wait List Control | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Customized [Mean (Full Range); unit: Years] — Adult individuals of any age were permitted, but since most of those diagnosed with cancer are older, the sample is predominantly older.
  Years
    Mean | 69.42 [55 to 84] | 69.42 [55 to 84] | 69.42 [55 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 10 | 12 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 10 | 11 | 21
  All other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient-Reported Outcomes Measurement System Scale, a Scale Developed by the National Institute of Health to Assess Outcomes Across Different Trials.
Description: The investigators will use the Patient-Reported Outcomes Measurement System which can be found on the National Institutes of Health website. It measures changes in scale levels of Depression, Anxiety, Fatigue, Sleep Disturbance before and after the intervention. The measure is developed by National Institutes of Health to permit comparison across studies, and is reliable and valid. This is measured at baseline, and to assess for change, after the 8 week yoga intervention. There are six items in each subscale with four points each, with a range from 1-5. The full subscale range is 6-30. Anxiety was assessed by anxiety subscale, ranging from 6 ( no anxiety) to 30 (worst possible anxiety); Insomnia was assessed by the anxiety subscale, ranging from 6 ( no anxiety) to 30 (worst possible anxiety).
Time Frame: Primary outcome is measured at baseline and after the 8 week yoga intervention.
Population: This is a small scale pilot study. Due to small sample size, we did pre-post analysis of the total groups, separated by those with and without initial impairment.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Pre Group Values: Patient Reported Outcome Measurement System values for all participants prior to participation in 8 session Yoga Therapy with home practice
- Post Group Values: Patient Reported Outcome Measurement System values for all participants after participation in 8 session Yoga Therapy with home practice
Arm/Group | Pre Group Values | Post Group Values
Number analyzed (Participants) | 23 | 23
units on a scale
  Anxiety within normal limits at start (n=18) | 8.90 [6 to 19] | 12.26 [6 to 24]
  Anxiety impaired at start (n=5) | 19.80 [17 to 24] | 16.80 [11 to 21]
  Insomnia within normal limits at start (n=16) | 12.41 [7 to 20] | 13.00 [6 to 30]
  Insomnia impaired at start (n=7) | 23.14 [21 to 30] | 18.14 [12 to 26]
Statistical Analysis 1: Comparison: Pre Group Values vs Post Group Values; Repeated measure Analysis of Variance (ANOVA) with null hypothesis of no group differences, comparing anxiety scores pre-Yoga versus post-Yoga, between the two groups for changes in anxiety; Test type: Superiority or Other; p = .004, ANOVA — The a priori threshold for statistical significance is .05. The .004 value exceeds this value. There was only one comparison, so there was no adjustment for multiple comparison. This analysis refers to the row and category of anxiety; F=10.25
Statistical Analysis 2: Comparison: Pre Group Values vs Post Group Values; Repeated measure Analysis of Variance (ANOVA) with null hypothesis of no group differences, comparing insomnia scores pre-Yoga versus post-Yoga, between the two groups. This measures changes in insomnia; Test type: Superiority or Other; p = .056, ANOVA — F=4.07. The a priori threshold for statistical significance is .05. The .056 value does not exceed it. There was only one comparison, so there was no adjustment for multiple comparison. This analysis refers to the row/category of insomnia

ADVERSE EVENTS:
Time Frame: We collected "serious adverse event and other (not including serious) adverse event" information from the beginning of the study period to 3 months post study period for a total of 5 months.
Description: During the collection period, two forms were submitted to the Institutional Review Board for review as required. One participant in the Arm 1, Yoga therapy, age 80, was hospitalized. His principal diagnosis was influenza. One participant in the Arm 2, Wait list, age 65, was hospitalized. His principal diagnosis was pneumonia.
Groups:
- Yoga Therapy: Received yoga therapy.
  One participant in the Arm 1, Yoga therapy, age 80, was hospitalized. His principal diagnosis was influenza.
- Wait List: Received no yoga therapy for 8 weeks while the intervention group received yoga therapy
  One participant in the Arm 2, Wait list, age 65, was hospitalized. His principal diagnosis was pneumonia.
- Wait List on Yoga Therapy: Received yoga therapy after an 8 week wait.
  No participants were hospitalized.
Arm/Group | Yoga Therapy | Wait List | Wait List on Yoga Therapy
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/11 | 1/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga Therapy (N=11) | Wait List (N=12) | Wait List on Yoga Therapy (N=12)
Influenza Unrelated Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — One participant in the Arm 1, Yoga therapy, age 80, was hospitalized for influenza. The reportable event is hospitalization, hence I am listing an Unrelated Hospitalization for Influenza.
Pneumonia Unrelated Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — One participant in the Arm 2, Wait list, age 65, was hospitalized for pneumonia. The reportable event is hospitalization, hence I am listing an Unrelated Hospitalization for Pneumonia

LIMITATIONS AND CAVEATS:
The goals of this study were modest. A small pilot pre-post randomized trial was completed with a Yoga therapy intervention and a Wait list intervention. Additional studies in larger samples are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes